CLINICAL TRIAL: NCT05026216
Title: To Assess the Effectiveness of Multiple Dose, Multiple Concentrations of Clostridium Histolyticum-aases, Qwo, for the Treatment of Mild to Moderate Cellulite in Adult Females to the Buttocks and Thighs
Brief Title: To Assess the Effectiveness of Multiple Dose, Multiple Concentrations of Qwo, for the Treatment of Mild to Moderate Cellulite.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: DMR Research, PLLC (Other)
Collaborators: Endo Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DMRR-001
Record Dates: First submitted 2021-03-26; First posted 2021-08-30 (Actual); Last update posted 2021-09-21 (Actual); Status verified 2021-09

CONDITIONS: Cellulite
MeSH Terms: conditions — Cellulite

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Single-arm study (Experimental): Using CCH-ases on bilateral buttocks and thigh injections. No placebo being used.
  Interventions: Drug: Qwo

INTERVENTIONS:
Drug: Qwo — Collagenase clostridium histolyticum-aaes is a combination of bacterial collagenases AUX-I and AUX-II, in an approximate 1:1 mass ratio, which are isolated and purified from the fermentation of Clostridium histolyticum bacteria. Collagenase AUX-I is a single polypeptide chain consisting of approximately 1000 amino acids. Collagenase AUX-II is a single polypeptide chain consisting of approximately 1000 amino acids.

SUMMARY:
This is a single center, off-label, multiple dose, multiple injection areas, Phase 4 study to assess the safety and efficacy of multi-dilution CCH in adult women with mild or moderate edematous fibrosclerotic panniculopathy (EFP). 5 subjects will be screened and dosed in the buttock and thigh areas using a multi-dilution injection technique.

Qualified subjects (determined by investigator assessment) will receive a single vial of 0.84 mg of CCH to treatment areas (buttocks and thighs) for a total dose of 1.68 mg in both buttocks and both thighs per treatment session × 3 treatment sessions (Day 1, Day 22, and Day 43). Subjects will have follow-up visits at approximately 90 after Day 1.

ELIGIBILITY:
Subject Inclusion Criteria:

In order to be eligible to participate in the study, at the Screening Visit and on Study Day 1, subjects must:

* Be female and 18-60 years of age at the time of consent.
* Have both buttocks and both posterolateral thighs with:

  * A score of 2 or 3 (mild or moderate) as reported by the investigator using the Clinician-Reported Photonumeric Cellulite Severity Scale (CR-PCSS).
  * A Hexsel Cellulite Severity Scale (CSS) Subsection D "Grade of Laxity, Flaccidity, or Sagging Skin" score of 0 (absence of laxity, flaccidity, or sagging skin), or 1 (slightly draped appearance) at the Screening Visit only.
* Have a body mass index (BMI) score between 18.0 kg/m2 and 30.0 kg/m2 and intends to maintain stable body weight (:S10% change from the Day 1 Visit weight) throughout the duration of the study (from the Screening Visit through the Day 180/Early Termination Visit).
* Be willing to apply sunscreen to the treatment areas before each exposure to the sun for the duration of the study (from the Screening Visit through the Day 180/Early Termination Visit).
* Be judged by the investigator to be in good health, based upon the results of a medical history and physical examination,.
* Be of nonchildbearing potential (history of hysterectomy, bilateral oophorectomy, bilateral tubal ligation, or postmenopausal with no history of menstrual flow in the 12 months prior to the Screening Visit); or, if of childbearing potential, be nonpregnant, nonlactating, and agree to use effective contraception when with a male partner for the duration of the study. Acceptable forms of contraception include hormonal measures (oral contraceptive pills, contraceptive patch, contraceptive ring, injections, etc), intrauterine devices, double barrier method (condom plus diaphragm, condom or diaphragm plus spermicidal gel or foam), surgical sterilization of the male partner, and abstinence.
* Have a negative serum pregnancy test at the Screening Visit and a negative urine pregnancy test prior to dosing at each treatment session.
* Be willing and able to comply with all protocol required visits and assessment Be able to read, understand, and independently complete patient reported outcome instruments in English.
* Be able to read, understand, and independently complete patient reported outcome instruments in English.
* Be adequately informed and understand the nature and risks of the study and be able to provide consent as outlined in Section 10.1.3.

Subject Exclusion Criteria

* A subject is ineligible for study participation if, at the Screening Visit or on Day 1, the subject:
* Is from a vulnerable population, as defined by the United States (US) Code of Federal Regulations (CFR) Title 45, Part 46, Section 46.111(b) and other local and national regulations, including but not limited to, employees (temporary, part-time, full-time, etc) or a family member of the research staff conducting the study, or of the sponsor, or of the contract research organization, or of the Institutional Review Board (IRB)/Independent Ethics Committee (IEC).
* Has a history of sensitivity or allergy to collagenase or any other excipient of CCH.
* Has any of the following systemic conditions:

  * Coagulation disorder.
  * Evidence or history of malignancy (other than excised basal-cell carcinoma) unless there had been no recurrence in at least 5 years.
  * History of keloidal scarring or abnormal wound healing.
  * Concurrent diseases or conditions that might interfere with the conduct of the study, confound the interpretation of the study results, or endanger the subject's well-being. Any questions about concurrent diseases will be discussed with the Medical Monitor.
  * Evidence of clinically significant abnormalities on physical examination.
* Has any of the following local conditions in the areas to be treated (both buttocks and both thighs):

  * History of lower extremity thrombosis or post-thrombosis syndrome.
  * Vascular disorder (eg, varicose veins, telangiectasia).
  * Inflammation or active infection.
  * Active cutaneous alteration including rash, eczema, or psoriasis.
  * A tattoo or other artificially inflicted body marker.
  * Has a mole located within 2 cm of any injection site.
* Has skin laxity or linear undulations on the treatment region (both buttocks or both thighs) that can be effaced by lifting skin.
* Has a Hexsel CSS Subsection D "Grade of laxity, flaccidity, or sagging skin" of 2 (moderate draped appearance) or 3 (severe draped appearance).
* Requires anticoagulant or antiplatelet medication during the study or has received anticoagulant or antiplatelet medication (except for :S150 mg aspirin daily) within 7 days before injection of study treatment.
* Has used any of the following for the treatment of EFP on either thigh and either buttock within the timelines identified below or intends to use any of the following at any time during the course of the study:

  * Liposuction during the 12-month period before dosing with study treatment.
  * Injections (eg, mesotherapy, dermal fillers, biostimulatory fillers); radiofrequency device treatments; laser treatment; buttock and thigh implant treatment; cryolipolysis; or surgery (including subcision and/or powered subcision) during the 12-month period before injection of study treatment.
* Any investigational treatment for EFP on a buttock and thigh during the 12-month period before the injection of study treatment.
* Endermologie or similar treatments during the 6 month period before injection of study treatment.
* Massage therapy during the 3-month period before injection of study treatment. Creams (eg, Celluvera™, TriLastin®) and/or home therapies to prevent or mitigate EFP during the 2-week period before injection of study treatment.
* Has received any collagenase treatments at any time prior to treatment in this study and/or has received previous treatment with EN3835 or CCH for cellulite.
* Has received treatment with an investigational product within 30 days (or 5 half-lives, whichever is longer) of the Screening Visit.
* Is pregnant and/or is providing breast milk or plans to become pregnant and/or to provide breast milk during the course of the study.
* Intends to initiate an intensive sport or exercise program during the study.
* Intends to initiate an intensive weight reduction program during the study.
* Has any other condition(s) that, in the investigator's opinion, might indicate the subject to be unsuitable for the study.

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 5 (Actual)
Dates: Start 2021-03-29 (Actual); Primary Completion 2021-08-15 (Actual); Study Completion 2021-08-31 (Actual)

PRIMARY OUTCOMES:
Improved score iGAIS | Day 1/Baseline and Day 90
  The proportion of subjects with changed (+1 or better) score on the Investigator Global Aesthetic Improvement Scale. (I-GAIS) for buttock and thigh from Day 1(baseline) to Day 90(final visit).

SECONDARY OUTCOMES:
BODY-Q- APPRAISAL OF CELLULITE Copyright©2019 Memorial Sloan-Kettering Cancer Center, New York, USA. All rights reserved. | Day1/Baseline to day 90/final visit
  Mean change from Day 1/Baseline in Body-Q Appraisal of Cellulite to day 90/final visit. On a scale of 1-4, 1 being 'extremely bothered, 2 'moderately bothered, 3 'a little bothered' and 4, not at all bothered. Post treatment, it is anticipated that subjects will see a decrease in cellulite, therefore, scoring higher (3-4s) of little to not at all bothered.
Dilution Matrix | Dilution matrix to be used at treatment visits - Day 1, Day 22 and Day 43.
  To generate calculations to determine a matrix of buttock and thigh injections possible from a single 1.84 mg vial

CONTACTS AND LOCATIONS:
Locations (1):
- DMR Research, PLLC, Westport, Connecticut, United States

DOCUMENTS (1):
  • Study Protocol (2020-12-15): https://cdn.clinicaltrials.gov/large-docs/16/NCT05026216/Prot_000.pdf